CLINICAL TRIAL: NCT02395744
Title: The Occlusion Perfusion Catheter for Optimal Delivery of Paclitaxel for the Prevention of Endovascular Restenosis - Below the Knee
Brief Title: The COPPER-B Trial
Acronym: COPPER-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horizons International Peripheral Group (Other)
Collaborators: Advanced Catheter Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPG-CLIN-2015-01
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Cardiovascular Diseases; Peripheral Vascular Disease; Arterial Occlusive Diseases; Peripheral Arterial Disease; Critical Limb Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Vascular Diseases; Arterial Occlusive Diseases; Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC Treatment (Experimental): Paclitaxel administration using the OPC for the prevention of restenosis in infrapopliteal de novo and restenotic lesions and occlusions using a novel catheter, the OPC. Subjects will be treated with the endovascular intervention selected by the treating physician in reference vessels ranging from 2mm to 4mm in diameter. Following the achievement of optimal interventional results (≤ 30 percent residual stenosis without stenting and without flow-limiting dissection) the OPC will be placed at the interventional treatment area and paclitaxel will be delivered to the treated segment.
  Interventions: Other: Paclitaxel administration using the OPC

INTERVENTIONS:
Other: Paclitaxel administration using the OPC

SUMMARY:
The purpose of the COPPER - B study is to assess the feasibility, safety, and initial efficacy of paclitaxel administration using the OPC for the prevention of restenosis in infrapopliteal de novo and restenotic lesions and occlusions using a novel catheter, the OPC.

ELIGIBILITY:
General Inclusion Criteria:

* Willing and able to provide informed consent and comply with all study requirements;
* Candidate for an infrapopliteal percutaneous intervention;
* Must be ≥ 18 years of age;
* Rutherford category 3-6;
* Willing and able to tolerate dual anti-platelet therapy (DAPT) for a minimum of one (1) month;
* Labwork within acceptable limits according to standard of care;
* INR < 2.0 if on warfarin or not on warfarin;
* Sheath size used for the interventional procedure 6F, 7F, or 8F.

General Exclusion Criteria:

* Life expectancy < one (1) year;
* Planned amputation prior to procedure;
* Pregnancy or nursing (a pregnancy test is required for all women of childbearing capabilities ≤ 7 days prior to the index procedure);
* Previous intervention of the target vessel with a drug eluting balloon, or drug delivery catheter;
* Acute limb ischemia;
* Known allergy to paclitaxel;
* Known hypersensitivity to other drugs manufactured in Cremophor® EL (polyoxyethylated castor oil; e.g. Drugs containing polyoxyethylated castor oil are drugs such as miconazole, cyclosporine injection, nelfinavir mesylate, saperconazole, tacrolimus, and xenaderm ointment);
* Known allergy to anticoagulants;
* Known TRUE acetylsalicylic acid (ASA) allergy;
* Use of glycoprotein (GP) IIb/IIIa inhibitors during the procedure visit within 30 days prior to the index procedure;
* Target lesion treated with a cryoplasty balloon at the time of the index procedure;
* Current enrollment in another investigational device or drug study;
* After obtaining informed consent, at any point up to introduction of the OPC, the investigator determines the study subject is not appropriate for the study;
* Hemorrhagic stroke within three (3) months;
* Renal failure or chronic kidney disease with GFR ≤30 ml/min or MDRD GFR ≤30 ml/min per 1.73 m2 (or serum creatinine ≥2.5 mg/L within 30 days of index procedure or patient is on dialysis);
* Prior vascular surgery of the index limb.

Angiographic Inclusion Criteria

* Reference vessel diameter (RVD) ≥ 2mm and ≤ 4mm;
* Single or multiple lesions in the infrapopliteal arteries (AT, PT, peroneal);
* If single lesion treatment, the minimum lesion length required is 2cm;
* Lesion location must in the area from the origin of the trifurcation vessel to the ankle (top of the talus bone);
* Minimum of one vessel run-off;
* Pre-intervention percent DS ≥ 70%;
* Target vessel reconstitutes at/above the ankle;
* Infrapopliteal treatment prior to infrapopliteal OPC treatment resulting in ≤ 30% residual stenosis;
* Infrapopliteal interventional treatment length is within the area of 1cm below the level of the knee joint to the malleolus, except in the case where an anomalous take-off of an infrapopliteal artery comes of at mid-knee joint.

Angiographic Exclusion Criteria

* Flow limiting dissection requiring stent placement;
* Post PTA residual stenosis > 30% as visualized by treating physician;
* Perforation requiring a covered stent;
* Lesion is above the trifurcation;
* In-stent restenosis in target vessel;
* Significant (≥ 50% DS) inflow lesion or occlusion left untreated in the ipsilateral Iliac, SFA, or popliteal artery proximal to the target lesion;
* Lesions in the target vessel not treated with the OPC;
* Visible thrombus in the target artery or proximal to the target artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Freedom from clinically driven target lesion revascularization (CD-TLR) | 6 months
Freedom from major adverse events (MAEs) | 6 months

SECONDARY OUTCOMES:
Device success | Index Procedure
Improvement in Rutherford category | 6 Months
Improvement in ABI | 6 months
Freedom from Target Vessel Revascularization | 6 Months
Improvement in wound healing | 6 months
Device or procedure related serious adverse events (SAEs) | 1 month
Treatment related anticipated adverse events (AEs) | 1, 3, and 6 months
Treatment related serious adverse events (SAEs) | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Bunch, MD, FACC, Principal Investigator — Cardiology Associates
Locations (4):
- United States (4):
  - Cardiology Associates, Fairhope, Alabama
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Michigan Outpatient Vascular Institute, Dearborn, Michigan
  - Cardiovascular Associates of East Texas, Tyler, Texas